CLINICAL TRIAL: NCT01041235
Title: A Phase I, Open-label, Dose-escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Intravenously Administered ATI-1123, a Liposomal Docetaxel Formulation, on an Every 3 Week Schedule, in Patients With Advanced Solid Tumors
Brief Title: Safety Study of a Liposomal Docetaxel Formulation in Patients With Solid Tumors Who Have Failed Previous Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azaya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI1123-101
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Solid Tumor; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Non-Small Cell Lung
Keywords: Solid Neoplasms; Carcinoma; Breast; Ovarian; Ovary; Pancreas; Pancreatic; Lung; NSCLC; Non Small Cell Lung; Prostate; Gastric; Head and Neck
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATI-1123 (Experimental)
  Interventions: Drug: ATI-1123 (active drug = docetaxel)

INTERVENTIONS:
Drug: ATI-1123 (active drug = docetaxel) — Dose escalation starting at 15 mg/m2 given once every 3 weeks via IV
  Other Names: ATI-1123; ATI1123; Docetaxel; Docetaxol; Taxotere

SUMMARY:
The purpose of this study is to determine the safety profile, including the maximum tolerated dose (MTD), of ATI-1123 a liposomal formulation of docetaxel, in the treatment of cancer patients with advanced solid tumors.

DETAILED DESCRIPTION:
The majority of advanced stage human cancers are fatal if not treated promptly and aggressively. Standard treatments include chemotherapy, radiation therapy and surgery. Docetaxel, the active ingredient in ATI-1123 and the FDA approved drug Taxotere, is a chemotherapy given by IV to patients to treat various types of cancers.

Docetaxel is a poorly water soluble semi-synthetic taxane analog commonly used in the treatment of a variety of solid tumors including non-small cell lung, prostate, breast, gastric and head and neck cancer. Because of its poor water solubility it is formulated with co-solvents that can potentially contribute to treatment related adverse events such as hypersensitivity. Current taxane formulations often complicate drug delivery and can alter both pharmacokinetic and toxicity profiles.

Results from nonclinical evaluations show that ATI-1123 retains the antineoplastic activity of docetaxel while removing the need for unwanted solvents like Tween 80. The administration of ATI-1123 versus other docetaxel chemotherapy formulations is expected to reduce hypersensitivity reactions (redness, swelling, itching at the infusion site), eliminate the requirement for premedications, have a broader therapeutic index, and enhance systemic docetaxel exposure.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign a written IRB-approved informed consent form.
* Have a histologically confirmed solid tumor.
* Have progressive disease following standard/approved chemotherapy or have no appropriate alternative therapy available.
* Have one or more tumors measurable or evaluable as outlined by modified RECIST or evaluable by CT or MRI scan.
* Have an ECOG performance status of ≤ 2.
* Have a life expectancy of at least 3 months.
* Be ≥ 18 years old.
* Have a negative pregnancy test (if female of childbearing potential)
* Demonstrate acceptable hepatic function:
* Bilirubin ≤ upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN
* Demonstrate acceptable renal function:
* Serum creatinine ≤ 1.5 x ULN, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (Calculated according to the Cockroft and Gault formula)
* Demonstrate acceptable hematologic status:
* Absolute neutrophil count ≥ 1500/mm3
* Platelet count ≥ 100,000/mm3 (measured within 72 hours prior to initial dose)
* Hemoglobin ≥ 9 g/dL
* Demonstrate acceptable coagulation status:
* PT or INR within 1.5x ULN
* PTT within 1.5x ULN
* Have recovered from prior treatments (eg, surgery, radiation, chemotherapy, investigational therapies) sufficiently prior to Day 1 so that, in the opinion of the Investigator and/or Medical Monitor, the protocol objectives would not be compromised.
* Agree to use an effective contraceptive method (hormonal or barrier method; or abstinence) for the duration of the study and for 30 days after the last dose (for men and women of child-producing potential).

Exclusion Criteria:

* Have New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months prior to Day 1, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG).
* Have a seizure disorder requiring anticonvulsant therapy.
* Have active CNS metastasis. Patients with a history of CNS metastases will be eligible if they have been treated and are stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on stable dose of steroids for ≥ 1 week prior to enrollment.
* Have severe, chronic obstructive pulmonary disease with hypoxemia.
* Have active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
* Are pregnant or nursing.
* Have undergone radiation therapy, surgery, chemotherapy, or investigational therapy within 28 days prior to study entry (6 weeks for nitrosoureas or Mitomycin C).
* Are unwilling or unable to comply with procedures required in this protocol.
* Have a known history of infection with HIV, hepatitis B, or hepatitis C.
* Have a serious nonmalignant disease that, in the opinion of the Investigator and/or the Medical Monitor, could compromise protocol objectives.
* Are currently receiving any other investigational agent.
* Have exhibited allergic reactions to docetaxel, or a similar structural compound, biological agent, or formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the (MTD) and (DLTs) of ATI-1123 administered every 3 weeks, over a range of doses in patients with advanced solid tumors. | Duration of study
To establish the dose recommended for future phase II studies with ATI-1123. | End of Study

SECONDARY OUTCOMES:
To establish the pharmacokinetics of intravenously administered ATI-1123. | Cycle 1 (various time points within the cycle)
To observe patients for any evidence of antitumor activity of ATI-1123 by objective radiographic assessment. | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Tolcher, MD, Principal Investigator — South Texas Accelerated Research Therapeutics (START); John Nemunaitis, MD, Principal Investigator — Mary Crowley Cancer Research Center; Jon M Rogers, MD, Study Chair — Azaya Therapeutics, Inc (Medical Monitor)
Locations (2):
- United States (2):
  - Mary Crowley Cancer Research Centers (MCCRC), Dallas, Texas
  - Cancer Therapy and Research Center (CTRC), San Antonio, Texas

REFERENCES:
- See also: Mary Crowley Medical Research Center website — http://www.marycrowley.org
- See also: Cancer Therapty and Research Center (CTRC) — http://www.uthscsa.edu